CLINICAL TRIAL: NCT01411982
Title: Role of PACAP in Increased Platelet Count and Aggregability in Childhood Nephrotic Syndrome
Brief Title: Role of PACAP in Nehprotic Syndrome
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, Dr Benedicte Eneman, Doctor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S52866
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Nephrotic Syndrome
Keywords: PACAP (pituitary adenylate cyclase-activating polypeptide); Nephrotic syndrome; Thrombosis; Platelets
MeSH Terms: conditions — Nephrotic Syndrome; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will identify the role of PACAP (pituitary adenylate cyclase-activating polypeptide) deficiency in patients with nephrotic syndrome. PACAP is a neuropeptide that has a putative role as an inhibitor of megakaryopoiesis and platelet function. Patients with nephrotic syndrome show decreased PACAP plasma levels, due to urinary loss. We hypothesize that in severe nephrotic syndrome, plasma deficiency of PACAP enhances megakaryopoiesis and causes blood platelet activation, which contribute to the increased rate of thromboembolic disease in these patients.

To test our hypothesis, the role of PACAP deficiency on pro-thrombotic state in patients with nephrotic syndrome will be studied using patient blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* New patient with nephrotic syndrome of patient during relapse of nephrotic syndrome
* Under 16 years old
* Treatment for nephrotic syndrome not yet started by first sample collection

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: New patients with nephrotic syndrome of patients during a relapse of nephrotic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
PACAP levels in plasma and urine | 3 test moments: at baseline during nephrotic syndrome before start of treatment; 4 weeks after start of remission; 4 weeks after stop of corticosteroid treatment. Estimated total time frame: 5 months

SECONDARY OUTCOMES:
Platelet count | 3 test moments: at baseline during nephrotic syndrome before start of treatment; 4 weeks after start of remission; 4 weeks after stop of corticosteroid treatment. Estimated total time frame: 5 months
Platelet aggregability | 3 test moments: at baseline during nephrotic syndrome before start of treatment; 4 weeks after start of remission; 4 weeks after stop of corticosteroid treatment. Estimated total time frame: 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatrics, UZ Leuven, Leuven, Vlaams-Brabant, Belgium